CLINICAL TRIAL: NCT07251907
Title: Structured Handoff Using Intelligent Framework for Transitions (SHIFT) Trial: A Randomized Controlled Trial of AI-Assisted End-of-Rotation Handoff Between Hospitalists
Brief Title: Structured Handoff Using Intelligent Framework for Transitions Trial
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHIFT Trial
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Electronic Medical Record; Transitions of Care; Physician Workflow; Artificial Intelligence (AI); Large Language Model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): The control arm will continue usual care without access to the AI drafting feature. Attendings will prepare handoffs themselves using current workflows within Carelign.
- LLM Tool (Experimental): The intervention arm will have access to an LLM-assisted draft generation feature within Carelign. This will generate a draft of the handoff, which the provider will then edit as necessary before finalizing.
  Interventions: Other: LLM tool to draft handoff

INTERVENTIONS:
Other: LLM tool to draft handoff — The intervention arm will have access to an LLM-assisted draft generation feature within Carelign. The feature will be accessed via a 'Draft Handoff' button in the attending handoff tab. The LLM is hosted in Penn's HIPAA-compliant environment and prompt engineering was performed through a series of handoff-specific iterative prompts with continuous quality assessments by the study team. In addition to the structured prompt, it will receive the most recent progress note from the primary team (or admission note, when no progress note is available), and the most recent specialty consult notes (within 72 hours of date of service). Generated drafts are editable; clinicians must review and finalize all content prior to sharing with their colleagues.
  Arms: LLM Tool

SUMMARY:
Inpatient general medicine attendings will be randomized to have an LLM feature turned on to provide a draft of an off-service handoff within Carelign (an EHR-adjacent provider communication tool). Providers who have access to this feature will be clearly instructed that if they use the LLM-generated draft, they must review and edit it as necessary before finalizing. The study will assess measures of documentation burden (as it relates to writing handoff) - including time spent writing handoff - and work exhaustion in both intervention and control groups.

DETAILED DESCRIPTION:
The Structured Handoff Using Intelligent Framework for Transitions (SHIFT) Trial is a pragmatic, parallel-group randomized controlled trial designed to evaluate whether an artificial intelligence (AI) tool integrated into the Carelign handoff platform can reduce documentation time and burden among inpatient hospitalists. The AI feature uses a large language model (LLM) tuned for clinical summarization to generate an editable draft of the end-of-rotation handoff. Hospitalists randomized to the intervention arm will have access to a "Draft Handoff" button within Carelign, which automatically generates a structured, editable handoff draft using data from recent notes in the electronic health record. Clinicians are required to review and edit all draft content before finalizing and sharing the handoff with colleagues. Providers in the control arm will continue using standard handoff workflows within Carelign without AI assistance.

The study will be conducted on general medicine services at the Hospital of the University of Pennsylvania (HUP) and Penn Presbyterian Medical Center (PPMC). Eligible participants include attending hospitalists scheduled for at least five consecutive days on service. Providers will be randomized 1:1 to the intervention or control arm, stratified by site and team. The study will enroll approximately 90 hospitalists contributing about 120 eligible rotations over a 12-week period. The primary outcome is total time (in minutes) spent drafting the end-of-rotation handoff, measured using automated Carelign audit logs. Secondary outcomes include documentation burden (modified NASA Task Load Index), work exhaustion (Stanford Professional Fulfillment Index), and self-reported drafting time. Exploratory measures include tool usability (Net Promoter Score), receiving provider ratings of handoff quality, and electronic health record (EHR) usage metrics (total and after-hours "pajama time").

The trial is unblinded and will be conducted under real-world conditions to maximize generalizability. Analyses will follow an intention-to-treat approach, using linear mixed-effects models with random intercepts for provider to account for repeated rotations. All data will be stored and analyzed in secure, HIPAA-compliant institutional environments. The study has received approval from the University of Pennsylvania Institutional Review Board and Penn Medicine's AI Governance Council.

ELIGIBILITY:
Inclusion Criteria:

* General medicine attending physicians at HUP (Medicine, Solid Oncology) or PPMC (Medicine) services.
* Scheduled for ≥5 consecutive days on service.

Exclusion Criteria:

- Jeopardy attendings and moonlighters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Time spent drafting end-of-rotation handoff | Over the last 3 days of a given rotation
  Time (minutes) spent drafting the entire end-of-rotation handoff, calculated from Carelign audit logs as the duration between first and last edit per patient (capped at 30 minutes per patient), summed per rotation.

SECONDARY OUTCOMES:
Documentation burden | Beginning (baseline) and end of study (3 months)
  Measured via the modified NASA-Task Load Index
Work exhaustion | Beginning (baseline) and end of the study (3 months)
  Measured via the Stanford professional fulfillment index
Total time spent drafting handoff | Last day of rotation (varies by schedule, typically day 5, 7, or 14 on service)
  Measured via first and last edits (overall) in Carelign on last day of rotation

OTHER OUTCOMES:
Incoming provider ratings of handoff quality | Within 3 days of rotation start
  Survey measures of clarity, accuracy, and usability of handoff (measured on a 5-point Likert scale, with higher being better)
Overall time spent on EHR | Last day of rotation (varies by schedule, typically day 5, 7, or 14 on service)
  Total and after-hours time in the EHR on the last day of service

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania and Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No